CLINICAL TRIAL: NCT06134154
Title: Safety and Efficacy of Carbon Dioxide Gas for Endoscopic Insufflation in Children
Brief Title: Safety and Efficacy of Carbon Dioxide Gas for Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chinenye Dike, Assistant Professor of Pediatrics, Division of Pediatric Gastroenterology, Hepatology and Nutrition, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-300011252
Record Dates: First submitted 2023-10-24; First posted 2023-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air (Placebo Comparator)
  Interventions: Other: Endoscopic insufflation gas
- Carbondioxide (Experimental)
  Interventions: Other: Endoscopic insufflation gas

INTERVENTIONS:
Other: Endoscopic insufflation gas — Carbon dioxide gas versus air for endoscopic insufflation

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of air versus carbon dioxide gas insufflation for endoscopy in children.

The main question[s] it aims to answer are:

•to determine safety of CO2 Assess patient comfort (abdominal pain, flatulence and bloating) with CO2 use when compared to air.

DETAILED DESCRIPTION:
In this study, children (6 months -18 years) undergoing all endoscopic procedures that includes an upper endoscopy including but not limited to Esophagogastroduodenoscopy (EGD/ upper endoscopy), EGD/ Colonoscopy, Endoscopic Retrograde Cholangiopancreatography (ERCP), Endoscopic ultrasound (EUS) e.t.c after appropriate consent, will be randomized 1:1 to either Air or CO2 gas for endoscopic insufflation. We will record demographics (name, age, sex, MRN, race/ethnicity), anthropometrics including weight, height/length, weight for length (WFL), WFL z score, BMI, BMI z score, indication/ reason for scope, other co-morbidities (other medical problems), personnel involved (faculty only, vs faculty + trainee), minute by minute end tidal CO2 levels, minute by minute minute ventilation levels, baseline blood pCO2, and blood pCO2 after each procedure. Pre and post procedure patient reported abdominal pain, bloating and flatulence. Pre and post procedure nurse assessed pain. Pre and post procedure vital signs. Patients will be randomized using a sealed envelope method by the endoscopy technician. Both patients and providers will be blinded to arm of enrollment.

ELIGIBILITY:
Inclusion Criteria:

- Infants and children 6 months to 18 years undergoing any upper endoscopy related procedure including but not limited to EGD/Colonoscopy, ERCP, EGD only, EUS, EGD with foreign body removal, Enteroscopy.

Exclusion Criteria:

* Patients with American Society of Anesthesiology (ASA) Physical Status Classification System of 4 and above
* Children with chronic lung disease,
* Children who are wards of the state will be excluded.
* Children needing language interpreting services that is not Spanish.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain | baseline/ pre-procedure to immediately after the procedure
  Rates of abdominal pain from pre-procedure to immediately after the procedure

SECONDARY OUTCOMES:
PCO2 level | baseline/ preprocedural to immediately after the procedure
  Incidence of elevated carbon dioxide level in the blood from pre-procedure to post -procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No